CLINICAL TRIAL: NCT04957966
Title: An Ecological Momentary Music Intervention for the Reduction of Stress in the Daily Life of Turkish Immigrant Women
Brief Title: Ecological Momentary Music Intervention for the Reduction of Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Urs Nater, Professor, University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMMI-T Pilot
Record Dates: First submitted 2021-06-18; First posted 2021-07-12 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Stress, Psychological; Stress, Physiological; Discrimination, Racial
Keywords: Ecological Momentary Intervention; Music; Stress reduction; Discrimination; Cortisol; Alpha-Amylase
MeSH Terms: conditions — Stress, Psychological; Racism

STUDY DESIGN:
Intervention Model Description: Intra-individually randomized design: Random assignment (50:50) to either the intervention condition or the control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music listening vs. No music listening (Experimental): Random assignment (50:50) of every participant to one of the following two conditions: Music listening after a stressful/discriminatory event (i.e., intervention condition) or no music listening after a stressful/discriminatory event (i.e., control condition).
  Interventions: Behavioral: self-selected relaxing music

INTERVENTIONS:
Behavioral: self-selected relaxing music — 20 minutes music listening

SUMMARY:
Ethnic discrimination is a prevalent problem in the European Union and other regions. In view of the significant negative impacts of discrimination on mental and physical health, it is of high relevance to counteract these negative effects and provide appropriate interventions. This study aims to investigate the feasibility and the effectiveness of a mobile-based intervention, delivering self-selected relaxing music to buffer biological (salivary cortisol, salivary alpha-amylase) and psychological (perceived stress, perceived ethnic discrimination) stress reactions in moments of acute stress and perceived ethnic discrimination in the everyday life of Turkish immigrant women (N=20, age range 18-65 years). An intra-individually randomized design will be used, i.e., participants will be instructed on a random basis to either listen to music (intervention event) or not (control event). The whole study period consists of 35 days with a baseline period (week 1), intervention period (week 2-4), and post period (week 5). To investigate the feasibility of the intervention, post-monitoring interviews will be conducted after the end of the whole study period.

DETAILED DESCRIPTION:
The experience of unfair treatment because of one's own ethnicity, i.e., ethnic discrimination, constitutes a complex stressor which triggers both physical and psychological stress reactions. In this regard, women may constitute a particularly vulnerable group, as they may be confronted with intersectional stigmata, i.e., both ethnicity-related and gender-related stigmata. Considering the resulting health impairments many people with migration background are confronted with, it is of great importance to provide interventions with the potential to minimize those negative consequences. Recognizing this necessity, an ecological momentary music intervention was developed in order to reduce psychological and biological (cortisol, alpha-amylase) stress levels due to perceived ethnic discrimination in everyday life. The primary aim of this study is to investigate the feasibility and the effectiveness of this mobile-based intervention.

It is hypothesized that listening to music after an event of acute stress and/or ethnic discrimination will result in stronger decreases in psychological (perceived stress, perceived ethnic discrimination), and biological (cortisol, alpha-amylase) stress levels compared to no music listening in everyday life (immediate effect). Further, it is expected that a decrease in diurnal psychological and biological stress levels will be observed throughout the study period (intermediate effect) and that participants will start to consume or increase their deliberate consumption of music after an event of acute stress and/or ethnic discrimination in their everyday life after the intervention (behavior change). In addition, it is hypothesized that the feasibility of the intervention will be confirmed by participants' self-reports of high usefulness of and satisfaction with the intervention as well as by a high usage rate.

The study design is as follows: Baseline period (week 1), intervention period (week 2 to 4), post period (week 5).

During the baseline and post period, psychological and biological stress fluctuations and perceived ethnic discrimination in daily life will be assessed. To this end, participants will be signaled three times a day (9:00 am, 2:00 pm, 7:00 pm) in order to answer questions on their momentary levels of stress, perceived discrimination, positive and negative affect, and their music-listening activities (time-contingent data entries). Additionally, whenever a stressful or discriminatory event occurs, participants are instructed to initiate a data entry by themselves in order to report their momentary levels of stress, perceived discrimination, positive and negative affect, and to answer questions on the current situation. To investigate activities after such self-initiated, event-contingent data entries, the app will signal the participants 20 (post 1) and 35 minutes (post 2) later for an additional data entry. As part of every time-contingent and event-contingent report, participants will provide a saliva sample in order to examine biological stress markers: salivary cortisol levels as index of hypothalamic-pituitary-adrenal axis (HPA axis) activity, salivary alpha-amylase as index of autonomic nervous system (ANS) activity.

A daily diary assessment will be conducted every evening at the same time. In this diary, participants will be asked about their current perceived stress, perceived discrimination, positive and negative affect, fatigue, coping strategies. Additionally, they will be asked whether discriminatory events had happened over the course of the day and if so, to describe the event(s). For this data entry, no saliva sample will be collected.

During the Intervention period (week 2 to 4), the sampling protocol will be the same as in baseline and post period (i.e., time-contingent data entries, daily diary assessment, self-initiated event-contingent data entries, post 1, post 2). Additionally, after every self-initiated event-contingent report, participants will be randomly assigned (50:50) to either the intervention event (listening to music for 20 minutes) or the control event (no music listening, continue the activity before the data entry). This approach constitutes an intra-individually randomized design.

To investigate the feasibility of the intervention, qualitative data from post-monitoring interviews will be gathered at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Turkish immigrants (1st or 2nd generation)
* Weekly ethnic discrimination (at least 2 discriminatory events per week; value of or above 104 on the Everyday Discrimination Scale)
* 18-65 years
* Sex: female

Exclusion Criteria:

* Insufficient proficiency of the German language
* Body mass index (BMI) above 30 kg/m2
* Mental disorders (i.e., current major depressive episode, lifetime psychosis or bipolar disorder, borderline personality disorder, eating disorder in the past 5 years, substance-induced disorder in the past 2 years)
* Chronic somatic diseases
* Medical conditions or medications known to affect endocrine or autonomic functioning
* Abuse of alcohol in the past 6 months
* Drug use in the past year, cannabis use in the past 14 days
* Pregnancy
* Breastfeeding
* Impaired hearing or absolute pitch

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Participants' self-reports on the integrability of the study into the daily life | after 5 weeks
  6 open-ended questions of semi-structured interviews on the integrability of the study into the daily life of the participants
Participants' self-reports on the perceived effectiveness of the intervention | after 5 weeks
  5 open-ended questions of semi-structured interviews on the perceived effectiveness of the intervention
Perceived burden regarding the intervention | after 5 weeks
  10 items of a self-developed questionnaire on perceived burden regarding the intervention (5-point Likert Scales, higher scores indicate greater levels of perceived burden)
Satisfaction with the intervention | after 5 weeks
  Combination of the following 10 items to measure participants' satisfaction with the intervention:
  * 6 items of a self-developed questionnaire on satisfaction with the intervention (5-point Likert Scales, higher scores indicate greater levels of satisfaction)
  * adaption of 4 items of a self-developed satisfaction questionnaire (Loo Gee, 2018; 5-point Likert Scales, higher scores indicated greater levels of satisfaction)
Usage Rate of the App | Across the 5-week study period
  Timestamped log-data of the app to determine usage rate by the participants (higher usage rate indicates a greater feasibility of the intervention)
Change in Subjective Stress Experience | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: after 20 minutes music listening/ not music listening; T2: 15 minutes after T1
  Momentary stress level: visual analogue scales (VAS; 0-100, higher scores indicate a greater level of momentary stress)
Change in Short-Term Neuroendocrine Stress: Hypothalamic-Pituitary-Adrenal Axis | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: after 20 minutes music listening/ not music listening; T2: 15 minutes after T1
  Biological Marker: Salivary Cortisol
Change in Short-Term Neuroendocrine Stress: Autonomic Nervous System | from baseline period (week 1) to post period (week 5); during the course of the intervention: T0: directly after a stressful/discriminatory event, T1: after 20 minutes music listening/ not music listening; T2: 15 minutes after T1
  Biological Marker: Salivary Alpha-Amylase

SECONDARY OUTCOMES:
Change in participants' behavior regarding music listening | change from baseline period (week 1) to post period (week 5)
  Occurrence of music listening after a stressful/discriminatory event (greater occurrence of music-listening indicates a better outcome)
Change in positive and negative affect | every evening in the daily diary assessment for 35 days
  PANAS (Positive Affect Negative Affect Scale) is a self-report questionnaire that consists of two scales to measure positive affect and negative affect, each scale consists of 10 items (5-point Likert Scales, for every scale higher scores indicate greater positive/negative affect)
Change in fatigue | every evening in the daily diary assessment for 35 days
  5 items (one of each scale) of the MFI (Multidimensional Fatigue Inventory), a self-report questionnaire consisting of 20 items that are assigned to 5 scales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation (5-point Likert Scales, higher scores on each subscale indicate greater levels of each subscale-specific type of fatigue)
Change in coping behavior | every evening in the daily diary assessment for 35 days
  5 items of the Brief-COPE (Coping Orientation to Problems Experienced), a self-report questionnaire that consists of 28 items to measure effective and ineffective ways of coping with stressful life events; one item of each subscale: active coping, use of emotional support, use of instrumental support, venting, religion; 5-point Likert-Scales with higher scores for each subscale indicating a greater level of the subscale-specific coping behavior)
Change in avoidance behavior regarding discriminatory events | every evening in the daily diary assessment for 35 days
  Combination of the following 4 items to measure change in avoidance behavior:
  * 3 items of the avoidance subscale of the CSI (Coping Strategy Indicator), a self-report questionnaire of situational coping that consists of 33 items with the subscales avoidance, problem solving, and seeking social support (5-point Likert-Scales with higher scores indicating greater levels of avoidance behavior)
  * one self-developed item to measure avoidance behavior, in particular the item measures if the person avoided situations and/or persons for fear of being discriminated against (5-point Likert-Scales with higher scores indicating greater levels of avoidance behavior)
Change in anticipation of discriminatory events | every evening in the daily diary assessment for 35 days
  3 items of the Racism-related Vigilance Scale, a 6-item scale to measure heightened vigilance regarding discriminatory events (5-point Likert-Scales with higher scores indicating greater levels of anticipation of discriminatory events)

CONTACTS AND LOCATIONS:
Overall Officials: Ricarda Nater-Mewes, Dr. Dr., Principal Investigator — University of Vienna; Urs Nater, PhD, Principal Investigator — University of Vienna
Locations (1):
- University of Vienna, Vienna, Austria